CLINICAL TRIAL: NCT02404077
Title: Use of Clonidine to Prevent Withdrawal Following Prolonged Dexmedetomidine Infusions
Status: Completed | Type: Observational
Sponsor: Joseph D. Tobias (Other)
Responsible Party: Sponsor-Investigator, Joseph D. Tobias, Chairman, Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB15-00256
Record Dates: First submitted 2015-03-24; First posted 2015-03-31 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Sedation
Keywords: Patients; undergoing; ICU
MeSH Terms: interventions — Clonidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Clonidine: Patients who received clonidine following prolonged dexmedetomidine infusions
  Interventions: Drug: Clonidine

INTERVENTIONS:
Drug: Clonidine

SUMMARY:
The investigators' clinical practice makes use of oral clonidine as a means of transitioning from intravenous dexmedetomidine following prolonged infusions (more than 3-5 days). Although this is common clinical practice, there is limited clinical data to demonstrate the efficacy of this technique and to provide clonidine dosing guidelines. The purpose of this study is to retrospectively review the investigators' experience with the use of oral clonidine to prevent withdrawal following the prolonged administration of dexmedetomidine.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received clonidine during the transition from dexmedetomidine.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ICU patients who have been on prolonged dexmedetomidine infusions.
Sampling Method: Non-Probability Sample
Enrollment: 712 (Actual)
Dates: Start 2015-04; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Evidence of withdrawal | Twice a day from the first day of taper of dexmedetomidine until 72 hrs. after the last dose
  Withdrawal is assessed using the Withdrawal Assessment Tool-1 (WAT-1). The 19-item assessment consists of (1) a review of the patient's record for the past 12 hours, (2) direct observation of the patient for 2 minutes, (3) patient assessment during a progressive stimulated exam routinely performed to assess level of consciousness at the beginning of each 12-hour shift, and finally (4) assessment of post-stimulus recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph D Tobias, MD, Principal Investigator — Nationwide Children's Hospital